CLINICAL TRIAL: NCT02433132
Title: Study of Ion Transport From Nasal Epithelial Cells Collected by Brushing (CCBN) in the Diagnosis of Atypical Forms of Cystic Fibrosis
Brief Title: Cystic Fibrosis Diagnosis by Analyzing Nasal Brushing
Acronym: MUCO-BROCC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P120913
Record Dates: First submitted 2015-04-29; First posted 2015-05-04 (Estimated); Last update posted 2017-09-28 (Actual); Status verified 2017-09

CONDITIONS: Cystic Fibrosis; Atypical Form of Cystic Fibrosis
Keywords: Cystic fibrosis; Adults; Atypical form; Nasal brushing; Epithelial cells; Ion transport
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Diagnostic test (Other): Diagnostic test will be perform on cell from nasal brushing
  Interventions: Other: Nasal brushing

INTERVENTIONS:
Other: Nasal brushing — The CCBN test is to evaluate the ion transport in the nasal epithelial cells taken from a subject by brushing the inferior turbinate with a mini-brush after local anesthesia. Analysis of ion transport is carried out ex vivo on the primary culture of nasal epithelial cells after brushing

SUMMARY:
The diagnosis of CF is currently based on the discovery of two CFTR gene mutations and / or a positive sweat test (> 60mmol / l). A significant number of patients with atypical cystic fibrosis (chronic sino-pulmonary disease with a single mutation in the CFTR gene and / or a test of the intermediate sweat between 30 and 60 mmol / l) undetected by these techniques are behind specialized care while irreversible lung damage is already existed. Currently, the measurement of nasal potential difference in vivo (DPN), which evaluates the transportation of chlorine in the nasal epithelium with an electrode, is proposed for the diagnosis of atypical forms. However DPN dependent nasal local conditions when analysing do not always offer the possibility of concluding the diagnosis of cystic fibrosis. It is necessary to develop new and more reliable diagnostic tests for the detection of cases of atypical cystic fibrosis. The authors propose to develop a new diagnostic technique based on the study of bioelectric properties of a preparation of nasal cells of the subject obtained by brushing and placed in primary culture (CCBN).

DETAILED DESCRIPTION:
Autosomal recessive, CF is caused by mutations in the CFTR gene whose nature determines the clinical expression and severity of the disease affecting mainly the respiratory, digestive and genital. Respiratory pathology is mainly responsible for the morbidity and mortality of patients with cystic fibrosis. CFTR, which is ion channel carrying chlorine, plays an essential role in respiratory disease through its involvement in the changes of surface liquid covering the respiratory epithelial cells.

Currently the measurement of nasal potential difference in vivo (DPN) can cause arguments electrophysiological diagnosis of cystic fibrosis (chlorine transport default) for patients with atypical form but can be rendered difficult or non-interpretable by the lack of cooperation of the patient (especially in the children who do not support the presence of the probe into the nose) or mostly due to poor local conditions related to infectious diseases rhino sinus of these patients.

It is necessary to develop new and more reliable diagnostic tests for the detection of cases of atypical cystic fibrosis. The study of ion transport from nasal epithelial cells collected by brushing (NBC) in the diagnosis of atypical forms of cystic fibrosis is tested in this trial as a new diagnostic test.

This research will focus on three groups:

1. Of patients with cystic fibrosis adults.
2. adult patients with atypical form
3. people who do not have cystic fibrosis

Depending on the patient group, there will be only one CCBN or CCBN and DPN or CCBN and DPN and genetic analysis to verify the absence of mutation.

ELIGIBILITY:
Inclusion Criteria:

* For patients with cystic fibrosis and those with atypical form:

  • Inclusion at least 30 days after a general or local infection of the upper airways
* For controls:

  • No history or Sino-pulmonary pathology and negative identification of mutations in the CFTR gene
* For all subjects involved in research:

  * Information and obtaining informed consent of the subjects.
  * Age ≥ 18 years
  * affiliation to a social security scheme or of such a regime

Exclusion Criteria:

* For all participants :

  * Taking a per os corticoids or topical corticosteroid treatment in the nose in the month preceding the nasal brushing or measurement of nasal potential difference
  * ORL surgical history of under 2 months
  * cauterization of the inferior turbinate of under 2 months
  * Hypersensitivity to local anesthetics of the amide (such as lidocaine) or with one of the components, including methyl parahydroxybenzoate contained in the excipient.
  * Porphyria.
  * Epilepsy not controlled by treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2015-03; Primary Completion 2018-07 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Quality of the CCBN test | 14 days after nasal brushing
  The primary endpoint is composite. The diagnostic quality of the test CCBN is the analysis of nasal epithelial cells:
  * in basal short-circuit current,
  * in amiloride-sensitive current corresponding to ENaC
  * cyclic AMP-dependent current corresponding to CFTR

SECONDARY OUTCOMES:
Nasal potential difference | 14 days after nasal brushing
  The nasal potential difference will be evaluated :
  * in basal,
  * after infusion of a solution of amiloride,
  * after infusion of a solution without amiloride chloride,
  * after infusion of a solution of amiloride and isoproterenol (agonist of cAMP).

CONTACTS AND LOCATIONS:
Overall Officials: Virginie Prulière-Escabasse, MD, PhD, Principal Investigator — Centre Hospitalier Intercommunal of Creteil
Locations (1):
- Centre Hospitalier Intercommunal de Créteil, Créteil, France